CLINICAL TRIAL: NCT06646744
Title: Safety Study About the mRNA Vaccines Against COVID-19 in Pediatric Patients (PEDIVACOV-HCSC)
Brief Title: Safety Study About the mRNA Vaccines Against COVID-19 in Children (PEDIVACOV-HCSC)
Acronym: PEDIVACOV-HCSC
Status: Completed | Type: Observational
Sponsor: Ana Belen Rivas Paterna (Other)
Responsible Party: Sponsor-Investigator, Ana Belen Rivas Paterna, designed by Principal Investigator, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Other Study IDs: PEDIVACOV-HCSC
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-01

CONDITIONS: COVID-19 Vaccine Adverse Reaction
Keywords: COVID19 vaccine; Pharmacovigilance; Drug-Related Side Effects and Adverse Reactions
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Vaccinated children: Children between 5 and 12 years old vaccinated with 2 doses of an approved mRNA vaccione against COVID-19.
  Interventions: Biological: mRNA COVID-19 vaccine

INTERVENTIONS:
Biological: mRNA COVID-19 vaccine — Children will be vaccinated according to standard local procedure

SUMMARY:
Drugs side effects in children need to be evaluated in a different way because of their constant growth and body changes.

The use of COVID-19 vaccines (mRNA vaccines) is worldwide spread as a safety measure against the pandemic.

Although clinical trials have shown that vaccines are safe in the general population, specific real-life monitoring is needed to address the special situation that applies to children.

DETAILED DESCRIPTION:
Drug-related side effects are an important health problem causing an increase in health costs. Most of the related research is focused on the adult population, therefore evidence in pediatric patients is scarse. This situation remains true in the clinical trials of the mRNA vaccines against COVID-19, with most studies suggesting the need of a greater follow up and specific research that address the pediatric population. Even though vaccines seem to be a safe and effective ways to protect the population against the COVID-19 pandemic, more information is needed regarding the safety profile for pediatrics in the short and long term.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes between 5 and 12 years old.
* Pediatric patients with data included in the Clinico San Carlos' Hospital available for consultation.
* Acceptance by the parents/legal guardians for the participation and follow up.

Exclusion Criteria:

* None

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All the pediatric patients (between 5-12 years old) vaccinated in the Clinico San Carlos' Hospital
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Incidence of vaccine side effects | 10 days, 1 month and 6 months after vaccination
  Incidence of vaccine side effects

SECONDARY OUTCOMES:
Vaccine side effects | 10 days, 1 month and 6 months after vaccination
  Clinical description of side effects that occurre during follow up
Time to vaccine side effect | 10 days, 1 month and 6 months after vaccination
  Clinical description of side effect according to the time of appearance
Causality of side effects | 10 days, 1 month and 6 months after vaccination
  Evaluation of the causality by using the modified Karch-Lasagna modified scale
Severity of side effects | 10 days, 1 month and 6 months after vaccination
  Evaluation of the severity using de Venulet criteria and the spanish pharmacovigilance system
Vaccine and drug interactions | 10 days, 1 month and 6 months after vaccination
  Evaluation of the possible interaction between the vaccines and regularly prescribed drugs
Vaccine reactogenicity | 10 days, 1 month and 6 months after vaccination
  Evaluation of the difference reactogenicity between the first and second vaccine dose by recording the side effect appearance after each dose.
Perceived quality of the vaccination system | 10 days, 1 month and 6 months after vaccination
  Evaluation of the parents perceived quality of the vaccination system

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion para Investigación Biomedica Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Galindo R, Chow H, Rongkavilit C. COVID-19 in Children: Clinical Manifestations and Pharmacologic Interventions Including Vaccine Trials. Pediatr Clin North Am. 2021 Oct;68(5):961-976. doi: 10.1016/j.pcl.2021.05.004. Epub 2021 May 18. PMID 34538306
- [Background] Belen Rivas A, Arruza L, Pacheco E, Portoles A, Diz J, Vargas E. Adverse drug reactions in neonates: a prospective study. Arch Dis Child. 2016 Apr;101(4):371-6. doi: 10.1136/archdischild-2015-309396. Epub 2016 Jan 27. PMID 26819267
- [Background] Vargas E, Terleira A, Hernando F, Perez E, Cordon C, Moreno A, Portoles A. Effect of adverse drug reactions on length of stay in surgical intensive care units. Crit Care Med. 2003 Mar;31(3):694-8. doi: 10.1097/01.CCM.0000049947.80131.ED. PMID 12626971
- [Background] Omer SB, Benjamin RM, Brewer NT, Buttenheim AM, Callaghan T, Caplan A, Carpiano RM, Clinton C, DiResta R, Elharake JA, Flowers LC, Galvani AP, Lakshmanan R, Maldonado YA, McFadden SM, Mello MM, Opel DJ, Reiss DR, Salmon DA, Schwartz JL, Sharfstein JM, Hotez PJ. Promoting COVID-19 vaccine acceptance: recommendations from the Lancet Commission on Vaccine Refusal, Acceptance, and Demand in the USA. Lancet. 2021 Dec 11;398(10317):2186-2192. doi: 10.1016/S0140-6736(21)02507-1. Epub 2021 Nov 15. PMID 34793741
- [Background] Luxi N, Giovanazzi A, Capuano A, Crisafulli S, Cutroneo PM, Fantini MP, Ferrajolo C, Moretti U, Poluzzi E, Raschi E, Ravaldi C, Reno C, Tuccori M, Vannacci A, Zanoni G, Trifiro G; Ilmiovaccino COVID19 collaborating group. COVID-19 Vaccination in Pregnancy, Paediatrics, Immunocompromised Patients, and Persons with History of Allergy or Prior SARS-CoV-2 Infection: Overview of Current Recommendations and Pre- and Post-Marketing Evidence for Vaccine Efficacy and Safety. Drug Saf. 2021 Dec;44(12):1247-1269. doi: 10.1007/s40264-021-01131-6. Epub 2021 Nov 5. PMID 34739716
- [Background] Yan Z, Yang M, Lai CL. COVID-19 Vaccinations: A Comprehensive Review of Their Safety and Efficacy in Special Populations. Vaccines (Basel). 2021 Sep 28;9(10):1097. doi: 10.3390/vaccines9101097. PMID 34696205
- [Background] Zheng YJ, Wang XC, Feng LZ, Xie ZD, Jiang Y, Lu G, Li XW, Jiang RM, Deng JK, Liu M, Xu BP, Wei Z, Liu G, Lu XX, Jin RM, Liu ZS, Shang YX, Shu SN, Bai Y, Lu M, Liu GH, Luo WJ, Cui YX, Ye LP, Lin LK, Zhao DC, Shen AD, Shao JB, Xiong LJ, Gao LW, Wang TY; China National Clinical Research Center for Respiratory Diseases; National Center for Children's Health, Beijing, China; Group of Respirology, Chinese Pediatric Society, Chinese Medical Association; Chinese Medical Doctor Association Committee on Respirology Pediatrics; China Medicine Education Association Committee on Pediatrics; Chinese Research Hospital Association Committee on Pediatrics; Chinese Non-government Medical Institutions Association Committee on Pediatrics; China Association of Traditional Chinese Medicine, Committee on Children's Health and Medicine Research; Zhao ZY, Yang YH, Shen KL. Expert consensus on COVID-19 vaccination in children. World J Pediatr. 2021 Oct;17(5):449-457. doi: 10.1007/s12519-021-00465-6. Epub 2021 Oct 7. No abstract available. PMID 34618327